CLINICAL TRIAL: NCT04239521
Title: The Epidemiology, Management, and the Associated Burden of Mental Health, Atopic and Autoimmune Conditions, and Common Infections in Alopecia Areata
Brief Title: The Epidemiology, Management, and the Associated Burden of Related Conditions in Alopecia Areata
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Collaborators: Pfizer (Industry); University of Surrey (Other); University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: P005
Record Dates: First submitted 2020-01-09; First posted 2020-01-27 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Alopecia Areata; Depressive Episode; Recurrent Depressive Disorder; Anxiety Disorders; Atopic Dermatitis; Allergic Rhinitis; Asthma; Crohn Disease; Ulcerative Colitis; Pernicious Anemia; Type 1 Diabetes; Hashimoto Thyroiditis; Graves Disease; Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis; Systemic Lupus Erythematosus; Polymyalgia Rheumatica; Sjogren's Syndrome; Psoriasis; Vitiligo; Multiple Sclerosis; Celiac Disease; Upper Respiratory Tract Infection; Influenza; Lower Resp Tract Infection; Acute Bronchitis; Pneumonia; Gastrointestinal Infection; Skin Infection; Urinary Tract Infections; Genital Infection; Herpes Zoster; Herpes Simplex; Infection; Infection Viral
Keywords: Alopecia areata; Common mental health conditions; Depression; Anxiety; Autoimmune disease; Atopic conditions; Epidemiology; Incidence; Prevalence; Infection
MeSH Terms: conditions — Alopecia Areata; Depressive Disorder; Anxiety Disorders; Dermatitis, Atopic; Rhinitis, Allergic; Asthma; Crohn Disease; Colitis, Ulcerative; Anemia, Pernicious; Diabetes Mellitus, Type 1; Hashimoto Disease; Graves Disease; Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing; Lupus Erythematosus, Systemic; Polymyalgia Rheumatica; Sjogren's Syndrome; Psoriasis; Vitiligo; Multiple Sclerosis; Celiac Disease; Respiratory Tract Infections; Influenza, Human; Bronchitis; Pneumonia; Cellulitis; Urinary Tract Infections; Herpes Zoster; Herpes Simplex; Infections; Virus Diseases; Depression; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with a confirmed diagnosis of Alopecia areata within the study period will be included as cases for analysis.
  Interventions: Other: Exposure of interest (studies 2 & 3).
- Controls: The control cohorts will be defined by matching cases with patients who have never been diagnosed with Alopecia areata either prior to or during the study period, by age and sex, at General Practice practice level.
  Interventions: Other: Exposure of interest (studies 2 & 3).

INTERVENTIONS:
Other: Exposure of interest (studies 2 & 3). — Common mental health conditions consist of depressive episodes, recurrent depressive disorder and anxiety disorder Atopic conditions consist of Atopic dermatitis, allergic rhinitis, asthma Autoimmune conditions consist of Crohn's disease, ulcerative colitis, Coeliac disease, Pernicious anaemia, Type 1 diabetes, Hashimoto's thyroiditis, Grave's disease, Rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, Systemic lupus erythematosus, polymyalgia rheumatica, Sjögren's syndrome, Psoriasis, vitiligo, Multiple sclerosis

SUMMARY:
This study series consists of four related studies and aims to explore and describe many important elements of alopecia areata over three key areas: (1) the current epidemiology of alopecia areata, (2) the prevalence and incidence of psychiatric co-morbidities in people with alopecia areata, (3) the prevalence and incidence of autoimmune and atopic conditions in people with alopecia areata, and (4) the incidence of common infections in people with alopecia areata.

DETAILED DESCRIPTION:
The overall purpose of the first study (Study 1) is to describe the epidemiology of Alopecia areata (AA) and to assess the current level of primary care service utilisation and management patterns associated with patients diagnosed with AA.

The overall purpose of the second study (study 2) is to assess the prevalence and incidence of mental health conditions (depressive episodes, recurrent depressive disorder and anxiety disorder) in adult patients diagnosed with AA relative to a control population of patients without a diagnosis of AA. In addition, the study will determine both the treatment, 'sick day' and unemployment burden. Treatment burden comprises that of medications and psychological interventions used to treat mental health conditions in adult patients diagnosed with Alopecia areata.

The overall purpose of the third study (Study 3) is to assess the prevalence and incidence of atopic and autoimmune conditions in adult patients diagnosed with AA relative to a control population of patients without AA.

The overall purpose of the fourth study (Study 4) is to assess the incidence of common infections in adult patients diagnosed with AA relative to a control population of patients without AA.

ELIGIBILITY:
Inclusion Criteria:

* Patients contributing to Royal College of General Practitioners Research and Surveillance Centre(RCGP RCS) primary care database between January 1, 2009 and December 31, 2018, will be eligible for inclusion.
* Only patients aged ≥18 will be eligible for studies 2 and 3.
* Only patients aged ≥ 18 and ≤ 65 will be included in the unemployment and sick day analysis (study 2)

Exclusion Criteria:

* People with the alternative non-AA diagnoses.
* People with AA diagnosis within 6 months of registration.
* People with less than 1 year of follow up available

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: These studies will use routinely collected and collated data from the Royal College of General Practitioners Research and Surveillance Centre database to provide a broadly representative sample of the population of England.
Sampling Method: Non-Probability Sample
Enrollment: 51955 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Study 1: The incidence of Alopecia Areata | Overall during 2009-2018 inclusive
  The incidence of Alopecia areata within the study cohort during the study period
Study 1: The incidence of Alopecia Areata stratified by sociodemographic factors | Overall during 2009-2018 inclusive
  This will comprise of the incidence of Alopecia Areata over the study period, by age group, gender, ethnicity, and Social Economic Status.
Study 1:The annual rate of primary care visits for people with Alopecia Areata. | Within one year of diagnosis of Alopecia Areata
  The annual rate of visits to primary care for any reason within one year of diagnosis.
Study 1: Secondary care dermatology service utilisation | Within one year of diagnosis of Alopecia Areata
  The percent of people reviewed in secondary care dermatology services within one year of diagnosis of Alopecia Areata
Study 2: The prevalence of common mental health conditions in adult patients diagnosed with Alopecia Areata at the time of diagnosis | At the time of diagnosis in all patients diagnosed with Alopecia Areata 2009-2018 inclusive
  Prevalence of common mental health conditions (depressive episodes, recurrent depressive disorder and anxiety disorder) in adult patients diagnosed with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 2: Describe the incidence of common mental health conditions in adult patients with Alopecia Areata | Within two years of diagnosis of Alopecia Areata
  Incidence of common mental health conditions (depressive episodes, recurrent depressive disorder and anxiety disorder) in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 2: Describe the mental health medication treatment burden of adult patients diagnosed with Alopecia Areata. | Within two years of diagnosis of Alopecia Areata
  This will comprise of the number of medications used to treat mental health conditions in patients diagnoses with Alopecia Areata. Antidepressant medication classes to be examined comprise; selective serotonin reuptake inhibitors and related medications (serotonin and norepinephrine reuptake inhibitors (SNRIs)), tricyclic antidepressants and related medications (tetracyclic antidepressant), and monoamine oxidase inhibitors. Anxiolytic medications to be examined comprise all benzodiazepines and other related medications indicated for use in anxiety states.
Study 2: Number of patients diagnosed with Alopecia Areata receiving mental health psychological intervention. | Within two years of diagnosis of Alopecia Areata
  This will comprise of the number of psychological interventions used to treat mental health conditions in patients diagnoses with Alopecia Areata. Psychological interventions comprise of counselling, Cognitive Behavioural Therapy, and psychotherapy.
Study 3: Describe the prevalence of atopic and autoimmune conditions in adult patients diagnosed with Alopecia Areata at the time of diagnosis | At the time of diagnosis in all patients diagnosed with Alopecia Areata 2009-2018 inclusive
  Prevalence of atopic and autoimmune conditions in adult patients diagnosed with Alopecia Areata in a contemporary real-world population at diagnosis compared with matched controls.
Study 3: Describe the incidence of atopic and autoimmune conditions in adult patients with Alopecia Areata. | Within five years of Alopecia Areata diagnosis
  Incidence of atopic and autoimmune conditions in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of a composite of common infections in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of a composite of any common infection (composite comprising a diagnosis of: upper and lower respiratory tract infection, pneumonia, acute bronchitis, influenza, skin infection, urinary tract infection, genital infections, gastrointestinal infection, herpes simplex and herpes zoster) in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of a composite of viral infections in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of a composite of any viral infection (composite comprising a diagnosis of: influenza, herpes simplex and herpes zoster infections, bronchitis, and any upper respiratory tract infections specifically coded as being viral) in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.

SECONDARY OUTCOMES:
Study 1: Adjusted incidence rate ratios of Alopecia Areata within England by geographic region. | Overall during 2009-2018 inclusive
  By region across England.
Study 2: Prevalence (percentage) of common mental health conditions (depressive episodes, recurrent depressive disorder and anxiety disorder), by socio-demographic factors, in adult patients diagnosed with Alopecia Areata. | At the time of diagnosis in all patients diagnosed with Alopecia Areata 2009-2018 inclusive
  By age group, gender, ethnicity, and Social Economic Status.
Study 2: Describe the burden of 'sick days' in adult patients diagnosed with Alopecia Areata relating to mental health conditions. | Within one year of diagnosis of Alopecia Areata
  Sick days will be indicated by the issuing of Med 3 certification from primary care (Statement of Fitness for Work) certification.
Study 2: Describe the prevalence of unemployment in adult patients diagnosed with Alopecia Areata. | Within one year of diagnosis of Alopecia Areata
  Unemployment will be identified using Read codes relating to unemployment recorded in the clinical record or the issuing of an Incapacity Benefit (IB113) or Employment and Support Allowance (ESA113) form.
Study 4: The incidence of upper respiratory tract infection in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of upper respiratory tract infection in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of lower respiratory tract infection in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of lower respiratory tract infection in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of influenza infection in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of influenza or influenza-like illness (where direct swab confirmed diagnosis is not performed) in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of acute bronchitis in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of acute bronchitis in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of pneumonia in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of pneumonia in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of gastrointestinal infection in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of gastrointestinal infection in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of stool confirmed gastrointestinal infection in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of gastrointestinal infection confirmed by stool culture or microscopy results (or other microbiological diagnosis confirmation) in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of skin infection in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of skin infection in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of urinary tract infection in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of urinary tract infection in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of genital infection in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of genital infection in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of herpes zoster infection in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of herpes zoster infection in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.
Study 4: The incidence of herpes simplex infection in adult patients with Alopecia Areata | Within five years of Alopecia Areata diagnosis
  Incidence of any recorded diagnosis of herpes simplex infection in adult patients with Alopecia Areata in a contemporary real-world population compared with matched controls.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGovern, MD, Study Director — Momentum Data
Locations (1):
- Momentum Data Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data is confidential but can be made available in an anonymised form to bone fide researchers subject to the required data protection training and other requirements. All data will remain behind a firewall and will only be available for access through a secured computer network.
Supporting Information: Study Protocol
Time Frame: There is no pre-specified time-frame for data availability; this will be considered on an individual basis for each request.
Access Criteria: As above

REFERENCES:
- [Derived] Macbeth AE, Holmes S, Harries M, Chiu WS, Tziotzios C, de Lusignan S, Messenger AG, Thompson AR. The associated burden of mental health conditions in alopecia areata: a population-based study in UK primary care. Br J Dermatol. 2022 Jul;187(1):73-81. doi: 10.1111/bjd.21055. Epub 2022 May 11. PMID 35157313
- [Derived] Harries M, Macbeth AE, Holmes S, Thompson AR, Chiu WS, Gallardo WR, Messenger AG, Tziotzios C, de Lusignan S. Epidemiology, management and the associated burden of mental health illness, atopic and autoimmune conditions, and common infections in alopecia areata: protocol for an observational study series. BMJ Open. 2021 Nov 16;11(11):e045718. doi: 10.1136/bmjopen-2020-045718. PMID 34785540